CLINICAL TRIAL: NCT02325050
Title: A Phase 1, Randomized, Placebo-Controlled, Observer-Blind Study to Evaluate the Safety, Tolerability and Immunogenicity of Heterologous and Homologous Prime-Boost Regimens Using MVA-BN-Filo® and Ad26.ZEBOV Administered in Different Doses, Sequences and Schedules in Healthy Adult Subjects
Brief Title: A Safety and Immunogenicity Study of Heterologous and Homologous Prime-Boost Ebola Vaccine Regimens in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR106479; VAC52150EBL1002 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: Healthy; Ebola viruses; Ebola Viral Disease (EVD); Filoviruses; monovalent vaccine; Human adenovirus serotype 26 (Ad26) expressing the Ebola virus Mayinga variant glycoprotein (Ad26.ZEBOV); Modified Vaccinia Virus Ankara - Bavarian Nordic (MVA-BN) Filo-vector; Safety; Immunogenicity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (10):
- Group 1 (Experimental): Participants will receive MVA-BN-Filo/ Ad26.ZEBOV (Day 1 /Day 15) or Placebo (Day 1/Day 15). Participants will receive Ad26.ZEBOV (5x10^10 vp) on Day 360.
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26. ZEBOV; Other: Placebo
- Group 2 (Experimental): Participants will receive MVA-BN-Filo/Ad26.ZEBOV (Day 1 /Day 29) or placebo (Day 1/Day 29). Participants will receive Ad26.ZEBOV (5x10^10 vp) on Day 360.
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26. ZEBOV; Other: Placebo
- Group 3 (Experimental): Participants will receive MVA-BN-Filo /Ad26.ZEBOV/ (Day 1/Day 57) or placebo (Day 1/Day 57). Participants will receive Ad26.ZEBOV (5x10^10 vp) on Day 360.
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26. ZEBOV; Other: Placebo
- Group 4 (Experimental): Participants will receive Ad26.ZEBOV/ MVA-BN-Filo (Day 1/Day 29) or placebo (Day 1/Day 29). Participants will receive Ad26.ZEBOV (5x10^10 vp) on Day 360.
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26. ZEBOV; Other: Placebo
- Group 5 (Experimental): Participants will receive MVA-BN-Filo (Day 1 and Day 15) or placebo (Day 1 and Day 15). Participants will receive Ad26.ZEBOV (5x10^10 vp) on Day 360.
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26. ZEBOV; Other: Placebo
- Group 6 (Experimental): Participants will receive Ad26.ZEBOV (Day 1 and Day 15) or placebo (Day 1 and Day 15). Participants will receive MVA-BN-Filo (1*10^8 TCID50) on Day 360.
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26. ZEBOV; Other: Placebo
- Group 7 (Experimental): Participants will receive Ad26.ZEBOV/ MVA-BN-Filo (Day 1/Day 15) or Placebo (Day 1/Day 15). Participants will receive Ad26.ZEBOV (5x10^10 vp) on Day 360.
  Interventions: Biological: Ad26. ZEBOV; Biological: MVA-BN-Filo; Other: Placebo
- Group 8 (Experimental): Participants will receive Ad26.ZEBOV/ MVA-BN-Filo (Day 1 /Day 29) or Placebo (Day 1/Day 29). Participants will receive Ad26.ZEBOV (1x10^11 vp) on Day 360.
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26. ZEBOV; Other: Placebo
- Group 9 (Experimental): Participants will receive MVA-BN-Filo/ Ad26.ZEBOV (Day 1 /Day 8) or Placebo (Day 1/Day 8).
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26. ZEBOV; Other: Placebo
- Group 10 (Experimental): Participants will receive MVA-BN-Filo/ Ad26.ZEBOV (Day 1 /Day 15) or Placebo (Day 1/Day 15).
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26. ZEBOV; Other: Placebo

INTERVENTIONS:
Biological: MVA-BN-Filo — One 0.5 milliliter (ml) intramuscular (IM) injection of 1*10^8, (50%Tissue Culture Infectious Dose [TCID50]).
  Arms: Group 1; Group 10; Group 2; Group 3; Group 4; Group 5; Group 6; Group 9
Biological: Ad26. ZEBOV — One 0.5 mL IM injection of 5*10^10 viral particles (vp).
  Arms: Group 1; Group 10; Group 2; Group 3; Group 4; Group 5; Group 6; Group 7; Group 9
Biological: MVA-BN-Filo — One 0.5 milliliter (ml) intramuscular (IM) injection of 4.4*10^8, (50%Tissue Culture Infectious Dose [TCID50]).
  Arms: Group 7; Group 8
Biological: Ad26. ZEBOV — One 0.5 mL IM injection of 1*10^11 viral particles (vp).
  Arms: Group 8
Other: Placebo — One 0.5 mL IM injection of 0.9% saline.

SUMMARY:
The purpose of this study is to test the safety and immunogenicity of MVA-BN-Filo and Ad26.ZEBOV as heterologous and homologous prime-boost vaccine regimens in healthy adult participants.

DETAILED DESCRIPTION:
This study consists of 3 parts: the first and third part with standard doses and the second part with higher doses. All parts are randomized, placebo-controlled, observer-blind to evaluate the safety, tolerability and immunogenicity of MVA-BN-Filo and Ad26.ZEBOV administered in different doses, sequences and schedules to healthy adult participants. The study consists of a screening period of up to 28 days, a vaccination period in which participants will be vaccinated at baseline (Day 1) followed by a boost on Day 15, 29, or 57, and third vaccine 1-year post-prime (3rd vaccination is optional for subjects in groups 1-8). The total duration of the study will be about 1 year for participants who wiil receive boost vaccine and about 3 months for participants who will receive placebo and 2 year for participants who will receive a 3rd dose. Safety will be monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy on the basis of physical examination, medical history, and the investigator's clinical judgment
* Have a body mass index (BMI) ≥18.5 and <35.0 kg/m2
* Women of childbearing potential must have a negative serum β-human chorionic gonadotropin pregnancy test at screening, a negative urine pregnancy test immediately prior to each study vaccine administration, and practice adequate birth control measures from 28 days before the prime vaccination until at least 3 months after the boost vaccination as specified in the study protocol. If not heterosexually active at screening, must agree to practice adequate birth control measures if they become heterosexually active during their participation in the study (from screening onwards until at least 3 months after the boost vaccination). Agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during participation in the study (from screening onwards until at least 3 months after the boost vaccination)
* Women of non-childbearing potential, defined as postmenopausal (>45 years of age with amenorrhea for ≥2 years or any age with amenorrhea for ≥6 months and serum follicle-stimulating hormone [FSH] >40 mIU/mL) or surgically sterile (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), are not required to use the birth control methods as specified in the study protocol
* A man who has not had a vasectomy and is sexually active with a woman of childbearing potential must agree to use a double-barrier method of birth control, such as either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository. In case the female partner is using an adequate method of birth control, a single-barrier method of birth control for the male subject is acceptable. Men must also agree not to donate sperm during their participation in the study (from screening onwards until at least 3 months after the boost vaccination)
* Must be available and willing to participate for the duration of the study visits and follow-up, provide verifiable identification, and have a means to be contacted

Exclusion Criteria:

* Has been vaccinated with a candidate Ebola vaccine
* Has been diagnosed with Ebola disease or exposed to Ebola including travel to West Africa in the last 12 months. West Africa includes but is not limited to the countries of Guinea, Liberia, Mali, and Sierra Leone. Participants who anticipate traveling to epidemic Ebola areas before the start of the long-term follow-up period will also be excluded from enrollment into the study
* Has received any Ad26- or MVA-based candidate vaccine in the past
* Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccines), including known allergy to egg or aminoglycosides
* A woman who is pregnant or breast-feeding, or planning to become pregnant while enrolled in the study or within 3 months after the boost vaccination
* History of diabetes mellitus type 1 or type 2, including cases controlled with diet alone; thyroidectomy, or thyroid disease requiring medication during the last 12 months; uncontrolled hypertension as defined in the study protocol; or, major psychiatric illness and/or substance abuse problems during the past 12 months that in the opinion of the investigator would preclude participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2015-07-02 (Actual); Study Completion 2017-05-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 21 days after the last vaccination (up to Day 381)
Number of participants with serious adverse events | Up to the end of long term follow-up (up to Day 720)
Number of participants with reactogenicity (ie, solicited local and systemic adverse events) | 1 week after each study vaccine administration

SECONDARY OUTCOMES:
Immune responses to the study vaccine regimens as measured by a virus neutralization assay | up to Day 720 (Group 1-8); Day 360 (Group 9, 10)
Immune responses to the study vaccine regimens as measured by an enzyme-linked immunosorbent assay (ELISA) | up to Day 720 (Group 1-8); Day 360 (Group 9, 10)
Immune responses to the study vaccine regimens as measured by an enzyme-linked immunospot (ELISpot) assay | up to Day 720 (Group 1-8); Day 360 (Group 9, 10)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (1):
- Rockville, Maryland, United States